CLINICAL TRIAL: NCT05103813
Title: Protective Effect of Beraprost Sodium Tablets on Coronary Microcirculation Function and Ventricular Remodeling After Reperfusion Therapy for Acute ST Segment Elevation Myocardial Infarction
Brief Title: Protective Effect of Beraprost Sodium Tablets on Reperfusion Therapy for Acute STEMI
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Beraprost Sodium treat STEMI
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2021-10

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — beraprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Beraprost Sodium Tablets (Experimental)
  Interventions: Drug: Beraprost Sodium Tablets

INTERVENTIONS:
Drug: Beraprost Sodium Tablets — Protective effect of Beraprost Sodium Tablets on coronary microcirculation function and ventricular remodeling after reperfusion therapy for acute ST segment elevation myocardial infarction

SUMMARY:
Protective effect of Beraprost Sodium Tablets on coronary microcirculation function and ventricular remodeling after reperfusion therapy for acute ST segment elevation myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* It meets the diagnostic criteria of acute ST segment elevation myocardial infarction: ischemic chest pain lasts for more than 30 minutes and can not be relieved by taking nitroglycerin; ST segment elevation of ECG with two or more adjacent leads, limb lead ≥ 1mm, chest lead ≥ 2mm; Or new left bundle branch block; The serum markers of myocardial necrosis increased at least twice the normal value
* Acute myocardial infarction was confirmed by coronary angiography
* The clinical and angiographic data were complete
* Direct PCI was performed within 12 hours after onset

Exclusion Criteria:

* Those who do not cooperate in the inspection, have poor compliance and cannot guarantee the completion of the test
* Conscious disorder, obvious intellectual disorder and mental disorder
* With metal foreign bodies, such as metal prosthesis, intraocular metal foreign bodies, intracranial aneurysm clamp, etc
* People with claustrophobia
* Had a history of myocardial infarction, PCI and coronary artery bypass grafting
* Factors affecting ST segment changes of ECG: complete left bundle branch block, preexcitation syndrome, pacemaker ECG, etc

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events | 1 weeks after baseline
  The incidence of mace after 1 week of treatment
Major Adverse Cardiovascular Events | 6 months after baseline
  The incidence of mace after 6 months of treatment
Major Adverse Cardiovascular Events | 1 year after baseline
  The incidence of mace after 1 year of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People' S Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No